CLINICAL TRIAL: NCT00614796
Title: A Study Evaluating the Effects of a Structured Lifestyle Intervention on Daily Physical Activity Level of COPD Patients in the First, Second and Third Echelon.
Brief Title: A Structured Lifestyle Intervention on Daily Physical Activity Level in COPD
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groningen Research Institute for Asthma and COPD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COACH; NL12651.042.06
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Lifestyle; Pedometer
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5 counseling meetings of 30 min in the first 3 months. In counseling, patients will be stimulated individually to enhance a physically active lifestyle.
  Interventions: Behavioral: Coach, using a stepcounter with exercise counseling
- 2 (No Intervention): daily physical activity is assessed at baseline, 3 months, 9 months and 15 months. No counseling.

INTERVENTIONS:
Behavioral: Coach, using a stepcounter with exercise counseling — 5 counseling meetings of 30 min in the first 3 months. In counseling, patients will be stimulated individually to enhance a physically active lifestyle.
  Other Names: COACH
  Arms: 1

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is increasing in the Netherlands. COPD is characterized by a deterioration of lung function, a lowering physical activity level and a low state of quality of life.

The aim of this randomized controlled study is to investigate the effects of a structured lifestyle program compared with usual care (in the first, second and third echelon) on the physical activity level of COPD patients.

150 COPD patients (GOLD I-IV) will be included, aged between 40 and 80 years. In each echelon 25 patients will participate in a structured lifestyle program and 25 patients will be treated with usual care.

In the structured lifestyle program, patients will be stimulated individually to enhance a physically active lifestyle. The primary outcome parameter is daily physical activity (steps/ day) assessed with a pedometer.

According to the study protocol patients in the experimental group and the control group participate in four measurement sessions distributed over 15 months. In each assessment a physical fitness test, lung function and questionnaires are taken. Patients of the experimental group participate in five individual counseling sessions and one telephonic counseling.

DETAILED DESCRIPTION:
Background of the study: Chronic Obstructive Pulmonary Disease (COPD) is increasing in the Netherlands. The incidence of COPD is about 2-3 per 1000 and the prevalence of 12-19 per 1000 patients in the Dutch primary health care. The World Health Organization (WHO) states that its prevalence in 2020 will be on the fourth rank of death and the fifth rank of causes of disability-adjusted life years lost worldwide. COPD is characterized by a deterioration of lung function, a lowering physical activity level and a low state of quality of life.

Objective of the study: The aim of the study is to investigate the effects of a structured lifestyle program (in the first, second and third echelon) on the physical activity level of COPD patients

Study design: It concerns a randomized controlled study. In this study a structured lifestyle program will be compared with usual care in the first, second and third echelon of the health care.

Study population: 150 COPD patients (GOLD I-IV) will be included, aged between 40 and 80 years. In each echelon 25 patients will participate in a structured lifestyle program and 25 patients will be treated with usual care.

Intervention: A structured lifestyle program, based on the COACH method, will be used. This method was developed by the Institute of Human Movement Sciences of the University of Groningen (RUG). Using COACH, patients will be stimulated individually to enhance a physically active lifestyle.

Primary study parameters/outcome of the study: Daily physical activity (steps/ day)

Secondary study parameters/outcome of the study: Personal characteristics, Body Mass Index, Fat Free Mass, lung function (FEV1), physical fitness (arm strength, leg strength, respiratory muscle strength, 6MWT), COPD related costs, ADL activities, type of activity, attitude towards physical activity, health status, physical fitness, psychological factors (self-efficacy, depression), quality of life, fatigue.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: According to the study protocol patients in the experimental group and the control group participate in five measurement sessions. In each assessment a physical fitness test, lung function, questionnaires is taken. Al participants wear a pedometer to registrate the number of steps a day during 2 weeks after each appointment. Patients of the experimental group participate in five individual counseling sessions and one telephonic counseling. As a result of the type of assessments used, the study has a very low risk profile.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years
* COPD GOLD stage I-IV
* Written informed consent

Exclusion Criteria:

* Comorbidity, like serious cardiovascular problems, serious limitations in neuromuscular performance and exacerbations in the previous two months, which can effect the outcome of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2006-11; Primary Completion 2009-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Daily physical activity in steps counts a day | Experimental group: assessment during first 3 months, 2 week assessment at 6 months, 9 months and 15 months. Control group: 2 weeks assessment at baseline, 3 months, 9 months and 15 months

SECONDARY OUTCOMES:
Personal characteristics | assessment at baseline
Body Mass Index | assessment at baseline, 3 months, 9 months and 15 months
Fat Free Mass | assessment at baseline, 3 months, 9 months and 15 months
Lung function (FEV1) | assessment at baseline, 3 months, 9 months and 15 months
Physical fitness (arm strength, leg strength, respiratory muscle strength, 6MWT) | assessment at baseline, 3 months, 9 months and 15 months
COPD related costs | assessment at 3 months, 9 months and 15 months
Type of activity, attitude towards physical activity, health status, physical fitness, psychological factors (self-efficacy, depression), quality of life, fatigue. | assessment at baseline, 3 months, 9 months and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Johan B Wempe, Phd, MD, Principal Investigator — University Medical Center Groningen
Locations (4):
- Netherlands (4):
  - Wilhelmina Ziekenhuis, Assen
  - Delfzicht ziekenhuis, Delfzijl
  - University Medical Centre Groningen, Groningen
  - Diaconessenhuis, Meppel

REFERENCES:
- [Derived] Altenburg WA, ten Hacken NH, Bossenbroek L, Kerstjens HA, de Greef MH, Wempe JB. Short- and long-term effects of a physical activity counselling programme in COPD: a randomized controlled trial. Respir Med. 2015 Jan;109(1):112-21. doi: 10.1016/j.rmed.2014.10.020. Epub 2014 Nov 22. PMID 25499548
- [Derived] Altenburg WA, Bossenbroek L, de Greef MH, Kerstjens HA, ten Hacken NH, Wempe JB. Functional and psychological variables both affect daily physical activity in COPD: a structural equations model. Respir Med. 2013 Nov;107(11):1740-7. doi: 10.1016/j.rmed.2013.06.002. Epub 2013 Jun 28. PMID 23810269